CLINICAL TRIAL: NCT04856878
Title: Effect of Single-dose Vancomycin After Catheter Replacement for Suspected Central Line-associated Bloodstream Infection (CLABSI) on Resolution of Infection in Critically Ill Patients: A Single Center Randomized Open Label Controlled Trial
Brief Title: Effect of Vancomycin After Catheter Replacement
Acronym: VanCat
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SD02
Record Dates: First submitted 2021-04-16; First posted 2021-04-23 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI); Catheter-related Bloodstream Infection
Keywords: Central Line-associated Bloodstream Infection; Catheter-related Bloodstream Infection; Vancomycin; Critical Care; Bloodstream Infection
MeSH Terms: conditions — Sepsis | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Standard of care (SOC) + single-dose intravenous vancomycin 15mg/kg
  Interventions: Drug: Vancomycin
- Control (No Intervention): Standard of care (SOC)

INTERVENTIONS:
Drug: Vancomycin — The investigational drug vancomycin is administered intravenously through a newly inserted peripheral or central venous catheter directly after removal of the 'old' catheters. The investigational drug is administered with a volume of 500ml normal saline (NaCl 0.9%) with a rate of maximal 1g per hour.
  Arms: Intervention

SUMMARY:
Randomized controlled trial of the effect of a single-dose intravenous Vancomycin after catheter replacement for suspected central line-associated bloodstream infection on resolution of infection in critically ill patients.

DETAILED DESCRIPTION:
Patients on the local intensive care unit with suspicion of central line-associated bloodstream infection will be randomized to standard of care consisting of catheter replacement and blood and catheter tip cultures and to standard of care plus a single-dose vancomycin. The effect of the intervention on resolution of humoral inflammation and negativity of blood cultures will be assessed after 48 and 96 hours.

ELIGIBILITY:
Inclusion Criteria:

Suspected central line-associated bloodstram infection defined as:

* Catheterization with a non-tunneled CVC and
* Clinical signs of local catheter infection or any increase in humoral inflammatory markers (PCT, CRP, WBC) or elevated body temperature ≥ 38.3°C not otherwise explained.

Baseline CRP at screening ≥ 100 mg/L

Exclusion Criteria:

* known positive blood cultures at the time of randomization
* High risk situation warranting immediate empiric antibiotic therapy:
* endovascular implant (prosthetic valve, pacemaker, vascular graft)
* high-risk for endocarditis warranting endocarditis-prophylaxis
* Septic shock
* Catheter replacement not feasible or no further indication for central venous catheterization
* Known hypersensitivity to vancomycin or any component of the formulation.
* Administration of Vancomycin, Teicoplanin, Daptomycin or Linezolid <48 hours before enrolment.
* Enrolment in another clinical study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of infection | 96 hours after catheter replacement
  Composite endpoint of absolute reduction of C-reactive protein and negativity of blood culture results at 48 and 96 hours (combinated with augmented binary method)

SECONDARY OUTCOMES:
Negativity of blood culture results | 48 hours and 96 hours after catheter replacement
  Negativity of blood culture results after 48 hours, 96 hours and both
Reduction of C-reactive protein | 48 hours and 96 hours after catheter replacement
  Absolute reduction of C-reactive protein (mg/dl) in plasma
Reduction of Procalcitonin | 48 hours and 96 hours after catheter replacement
  Absolute reduction of Procalcitonin (mcg/L) in plasma
Reduction of IL-6 | 48 hours and 96 hours after catheter replacement
  Absolute reduction of IL-6 (ng/L) in plasma
Reduction of white blood cell count | 48 hours and 96 hours after catheter replacement
  Absolute reduction of white blood cell count (G/L)
28-day survival | 28 days
  Survival after a follow-up of 28 days or until hospital discharge
ICU-free days at day 28 | 28 days
  Cumulative days not admitted to the intensive care unit in patients alive at day 28
Vasopressor-free days at day 28 | 28 days
  Cumulative days of no vasopressor therapy in patients alive at day 28
Invasive mechanical ventilation-free days at day 28 | 28 days
  Cumulative days of no invasive mechanical ventilation in patients alive at day 28
Antibiotic-free days at day 28 | 28 days
  Cumulative days of no antibiotic therapy in patients alive at day 28

OTHER OUTCOMES:
Incidence of central line-associated bloodstream infections | from blood cultures drawn before replacement and at 48 and 96 hours
  Definition according to the National Healthcare Safety Network (NHSN - CDC) Patient Safety Component Manual 2021
Blood culture | from blood cultures drawn before replacement and at 48 and 96 hours
  positivity of blood cultures
Vancomycin level in plasma | 24 hours after administration
  Vancomycin level (mg/L) in plasma after 24 hours
Incidence of acute kidney injury | 28 days
  Incidence of new or worsening acute kidney injury according to the definition and classification of the KDIGO 2012 guidelines
Hypersensitivity reaction to Vancomycin | 6 hours after catheter replacement
  Hypersensitivity reaction in the following 6 hours after vancomycin administration/catether replacement. Hypersensitivity reaction is defined as any new of the following symptoms: flushing, erythema, pruritus, pains or muscle spasms in the back or chest, dyspnea or hypotension.